CLINICAL TRIAL: NCT07134413
Title: Efficacy and Safety of QL1706 and Bevacizumab With or Without Chemotherapy in Patients With Non-Squamous Non-Small Cell Lung Cancer Previously Treated With Immune Checkpoint Inhibitors
Brief Title: QL1706/Bevacizumab ± Chemotherapy in Post-ICI Non-Squamous NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-NSCLC-QIBA-1002/CTONG2502
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: NSCLC
Keywords: iparomlimab and tuvonralimab; QL1706; Checkpoint inhibitor; NSCLC
MeSH Terms: interventions — Bevacizumab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706 plus bevacizumab combined chemotherapy (Experimental): Patients will receive QL1706 (5 mg/kg) plus bevacizumab (15 mg/kg) and chemotherapy (nab-paclitaxel, pemetrexed, or docetaxel) every 3 weeks.
  Interventions: Drug: QL1706 plus bevacizumab with or without chemotherapy
- QL1706 combined bevacizumab (Experimental): Patients will receive QL1706 (5 mg/kg) plus bevacizumab (15 mg/kg) every 3 weeks.
  Interventions: Drug: QL1706 plus bevacizumab with or without chemotherapy

INTERVENTIONS:
Drug: QL1706 plus bevacizumab with or without chemotherapy — QL1706(iparomlimab and Tuvonralimab) was generated by using MabPair, a new technological platform that enables the production of two antibodies close to their natural forms from a single host cell line and is manufactured as one product. QL1706 contains a mixture of anti-PD-1 IgG4 and anti-CTLA-4 IgG1 that were produced together in a fixed ratio. Each antibody was individually optimized to achieve desirable target coverage and antibody effector functions.
  Bevacizumab is a monoclonal antibody medication used to treat various cancers and a specific eye disease. It works by blocking a protein called VEGF, which helps tumors form new blood vessels, thus starving the tumor of nutrients and oxygen.
  Chemotherapy (nab-paclitaxel, pemetrexed, or docetaxel) Nab-paclitaxel, also known as nanoparticle albumin-bound paclitaxel, is a chemotherapy drug used to treat certain cancers. It's a form of paclitaxel that's bound to albumin nanoparticles, which improves its solubility and delivery to cance

SUMMARY:
The goal of this clinical trial is to evaluate QL1706 plus bevacizumab with or without chemotherapy in patients with PD-L1-negative, locally advanced or metastatic non-squamous non-small cell lung cancer (NSCLC) previously treated with immune checkpoint inhibitors (ICIs). The primary objectives are:

To assess the efficacy and safety of QL1706 combined with bevacizumab (± chemotherapy) in this population.

Eligible patients with PD-L1-negative, locally advanced or metastatic non-squamous NSCLC who progressed after prior PD-1/PD-L1 inhibitor therapy will be assigned to one of two treatment arms at the investigator's discretion:

Arm 1: QL1706 + bevacizumab + chemotherapy (target enrollment: 67 subjects). Single-agent chemotherapy (selected from regimens not previously received) will be administered, with options including nab-paclitaxel, pemetrexed, or docetaxel.

Arm 2: QL1706 + bevacizumab (target enrollment: 10 subjects).

ELIGIBILITY:
Inclusion Criteria:

1. Signed an informed consent form
2. Patients aged ≥18
3. Histologically or cytologically confirmed stage III or IV non-squamous non-small cell lung cancer (NSCLC) per the American Joint Committee on Cancer (AJCC) 8th Edition staging system
4. at least one measurable lesion according to RECIST 1.1 criteria
5. ECOG PS 0-1.
6. Subjects must have adequately documented disease progression following prior treatment with PD-1/PD-L1 inhibitors (administered as monotherapy or in combination with chemotherapy)

8. The most recent tumor tissue sample prior to the first dose of the study drug demonstrated PD-L1 TPS <1% 9. appropriate organ function

Exclusion Criteria:

1. Known presence of sensitizing mutations in EGFR, EGFR exon 20 insertions, ALK fusions, ROS1 fusions, RET fusions, NTRK fusions, BRAF V600E mutations, MET exon 14 skipping mutations, or HER2 sensitizing mutations (for other genetic alterations, eligibility will be determined by the Biomarker Committee on a case-by-case basis).
2. Patients with symptomatic, neurologically unstable central nervous system (CNS) metastases, or CNS diseases that require increased steroid doses to control
3. Prior lines of systemic anti-tumor therapy ≥ 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 2 years
  ORR is defined as the proportion of subjects with confirmed best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  From the first treatment to the date of first documentation of disease progression, or death due to any cause
Overall survival | 2 years
  From the first administration to death from any cause